CLINICAL TRIAL: NCT00856999
Title: Botox Cosmetic and the Young Patient With Glabellar Furrows
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Roger Dailey, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGNR-08-0093
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Glabellar Furrows
Keywords: Glabellar lines of moderate severity at maximum frown
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botox (Experimental): Botox Cosmetic will be delivered in standard doses of 4 units per injection site over a total of 5 sites, thus treating the procerus and corrugator superciliaris muscle groups
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — Botox Cosmetic will be delivered in standard doses of 4 units per injection site over a total of 5 sites, thus treating the procerus and corrugator superciliaris muscle groups

SUMMARY:
The purpose of this study is to see if consistent treatment with Botox will lead to longer lasting effects. Botox is an injectable liquid that is approved by the U.S. Food and Drug Administration to reduce wrinkles on the forehead in the area between the eyebrows. In this study a different dosing schedule of Botox injections will be used to see if the effects of the Botox treatment last longer than the effects of the standard injection regimen.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Fitzpatrick Skin Types I-III
* Between 30 and 50 years of age
* At least moderate severity at maximum frown

Exclusion Criteria:

* Prior botulinum toxin treatment
* Any disorder (such as myasthenia gravis, Eaton-Lambert syndrome) or agent (such as aminoglycoside antibiotics) that might interfere with neuromuscular function
* Any other condition or situation that might put the subject at significant risk, confound the study results (such as significant pre-existing brow or eyelid ptosis)
* Allergy or sensitivity to any study component
* Participation in another clinical study within 30 days of the study start date
* Are planning other facial cosmetic procedures during the study period, or are pregnant, breastfeeding, or planning a pregnancy during the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-02-08 (Actual); Primary Completion 2010-11-17 (Actual); Study Completion 2010-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Dailey, MD, Principal Investigator — Oregon Health and Science University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from medical practice and IRB approved media placement
Period: Overall Study
Arm/Group | Botox
Started | 50
Completed | 45
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Botox
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50
Facial wrinkle scale [Mean (Full Range); unit: units on a scale] — Four-point validated facial wrinkle scale (FWS) Minimum score = 0 (no wrinkles) Maximum score = 3 (deep wrinkles)
  units on a scale | 2.78 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Facial Wrinkle Scale
Description: Four-point validated facial wrinkle scale (FWS) Minimum score = 0 (no wrinkles) Maximum score = 3 (deep wrinkles)
  Baseline to 20 months is the active injection phase 20 months to 26 months is the follow-up phase
Time Frame: 26 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment: 26-month 2-phase study enrolling 50 toxin-naïve females aged 30-50 years with Fitzpatrick Skin Types I to III and moderate (2) to severe (3) glabellar lines on the 4-point Facial Wrinkle Scale at maximum contraction.
Arm/Group | Treatment
Number analyzed (Participants) | 50
units on a scale
  Physician Rating | 1.86 (0.65)
  Subject Rating | 2.10 (0.67)
Statistical Analysis 1: Comparison: Treatment; Test type: Equivalence — Non-parametric test equivalent to the dependent t-test; p < .001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Patient Assessed Frown-line Improvement
Description: Four-point satisfaction scale Neutral = 0 (minimum score) Somewhat satisfied = 1 Definitely satisfied = 2 Greatly satisfied = 3 Couldn't be more satisfied = 4 (maximum score)
  Baseline to 20 months is the active injection phase 20 months to 26 months is the follow-up phase
Time Frame: 20 months
Measure: Number; unit: percentage of patients
Groups:
- Treatment: Frown-line assessments
Arm/Group | Treatment
Number analyzed (Participants) | 50
percentage of patients
  Score 0 | 7
  Score 1 to 2.5 | 24
  Score 3 to 4 | 69
Statistical Analysis 1: Comparison: Treatment; Test type: Equivalence — Non-parametric test equivalent to the dependent t-test; p < .0004, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Botox
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No